CLINICAL TRIAL: NCT01999712
Title: Right Ventricular Failure After Implantation of Left Ventricular Assist Devices
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Kunal Bhatt, Assistant Professor, Emory University
Other Study IDs: IRB00058588; 13SDG15960001 (Other: Other)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure
Keywords: heart failure; left ventricular assist device; right ventricular failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma will be stored for biomarkers analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LVAD recipients: Patients who are scheduled for LVAD implantation will undergo preoperative echocardiography
  Interventions: Procedure: Echocardiography

INTERVENTIONS:
Procedure: Echocardiography — Patients will undergo an echocardiogram at baseline (preoperative) and at 30 and 90 days after LVAD implantation

SUMMARY:
The left ventricular assist device (LVAD) is a portable mechanical pump that helps the left side of the heart of patients with severe heart failure that are awaiting heart transplantation or are not transplant candidates. However, while LVAD supports the left side of the heart, the right side must work on its own. Sometimes the right side does not recover, a condition called right ventricular failure (RVF). This complication increases mortality, prolongs hospitalization, requires additional procedures, and increases costs. Several risk factors and scores have been proposed to identify patients at risk for RVF. However, these methods have proven inadequate; one out of three patients is still experiencing right ventricular failure after LVAD surgery.

Echocardiography, an established noninvasive method to see the heart without radiation or risk, has a lot of potential to identify patients at risk for RVF. The questions we will tray to answer with this American Heart Association funded project are:

1. Can echocardiography before scheduled LVAD surgery predict who is going to develop RVF and poor quality of life so we can better select patients for LVAD surgery?
2. Can echocardiography before scheduled LVAD surgery tell us the course of right ventricular function after implantation so we can potentially take additional measures and prevent RVF?

To answer these questions, we will record images of the heart with echocardiography before LVAD surgery in 120 LVAD recipients at Emory University. We will then follow the patients for 90 days to detect any symptoms and signs of clinical RVF and poor quality of life and record the course of right ventricular function with echocardiography.

Currently, it is estimated that 150,000 to 250,000 patients in US are potential LVAD recipients with 2,000 devices implanted in 2012. LVAD can improve survival and quality of life in suitable patients. However, implantation requires a major surgical procedure with associated risks and considerable resources. Thus, careful patient selection is necessary to minimize risk for patients and maximize benefit for patients and society. Our long-term goal is to use echocardiography as a tool to (1) optimally select patients for LVAD and offer alternatives to patients at increased risk for complications and (2) potentially, inform earlier LVAD implantation in patients with weakening right ventricular function.

DETAILED DESCRIPTION:
Despite (1) improved outcomes and lower rates of right ventricular failure (RVF) with the newer, continuous-flow left ventricular assist devices (LVAD) over pulsatile-flow devices and (2) development of clinical prediction scores to identify patients at risk for RVF post LVAD, RVF still occurs in 20% to 40% of recipients, even with the newer devices.

In 2012, 2000 LVADs were implanted in U.S. and the number is rapidly increasing. Post-LVAD outcomes depend critically on right ventricular (RV) function. RVF can lead to:

* Reduced survival and progression to transplant (Tx) and worse post-Tx outcomes
* Significantly higher rates of resources utilization
* Long-term poor exercise capacity and quality of life (QoL)

True echocardiographic quantification of RV function has only recently been considered in RVF prediction post LVAD; however these studies were retrospective and had inconsistent population and outcome definitions. Also, despite promising results in a retrospective study, preoperative RV mechanics have not been prospectively evaluated as RVF predictors to date.

In this study, we plan to enroll a total of 120 LVAD candidates to evaluate standard and mechanics-based echocardiographic measures of RV function for prediction of (1) RVF within 90 days; (2) QoL at 90 days; and (3) RV recovery at 90 days post LVAD implantation.

Aim 1: We will perform echocardiography within 7 days of planned LVAD surgery to evaluate the association of prespecified RV parameters with (1) RVF within 90 days and (2) QoL at 90 days. Our main hypotheses is an RV echo score will predict RVF within 90 days post LVAD with clinically relevant discrimination (C>0.85) and positive and negative predictive values (>80%). Our secondary hypothesis is that the RV score will predict poor QoL at 90 days with clinically relevant discrimination and predictive values.

Aim 2: We will repeat echocardiograms at 30 and 90 days post LVAD surgery to examine the association of baseline RV function with RV recovery. Our hypothesis is that the RV score will predict RV function recovery post LVAD and that RV mechanics will have incremental value for prediction of these outcomes.

These results may help improve LVAD outcomes and reduce resource utilization by facilitating shared decision-making and selection for LVAD vs. alternatives; provide insights into RV function recovery; and inform reassessment of LVAD timing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) Class 2-7
* Willing to participate
* Able to give consent

Exclusion Criteria:

* INTERMACS Class 1
* Pre-operative advanced RVF, defined as planned or anticipated need for RVAD or extracorporeal membrane oxygenation at surgery
* Unresponsive pulmonary vascular resistance (PVR) >6 Wood units

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for LVAD implantation seen at Emory University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Right ventricular failure | 90 days
  Right ventricular failure (RVF) at 90 days, defined as RVF-related death (multi-organ failure), need for inhaled nitric oxide postoperatively for ≥48h, need for post-operative inotropes for ≥14 days, reinstitution of inotropes beyond 14 days, or need for a RV assist device (RVAD)

SECONDARY OUTCOMES:
Quality of life | 90 days
  QoL by Kansas City Cardiomyopathy Questionnaire at 90 days defined as summary score <45
Right ventricular recovery | 30 and 90 days
  RV recovery, defined as 5% improvement in RV fractional area change at 30 days and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Andreas P Kalogeropoulos, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States